CLINICAL TRIAL: NCT01949012
Title: A Randomised Control Trial to Determine Whether Intervention Based on a Microstream Capnography-based Ventilation Monitoring System Will Decrease Hypoxaemaia During Intravenous Sedation With Midazolam.
Brief Title: Capnography Monitoring During Intravenous Conscious Sedation Sedation With Midazolam for Oral Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Cork (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Principal Investigator, Dr Paul Brady, Clinical Fellow, University College Cork
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Dental capnog
Record Dates: First submitted 2013-09-09; First posted 2013-09-24 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2015-05

CONDITIONS: Hypoxemia
Keywords: Midazolam; Endtidal carbon dioxide; Desaturation
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Standard monitoring
- Capnography (Experimental): Standard monitoring and capnography
  Interventions: Other: Capnography

INTERVENTIONS:
Other: Capnography — Capnography waveform and capnometry readings
  Arms: Capnography

SUMMARY:
Dentists use sedation to help patients accept difficult procedures and to relieve anxiety. During sedation, the well-being of the patient is monitored by the dental team. When carried out according to recognised guidelines,intravenous dental sedation is considered to be very safe. For some patients, dental sedation is a useful alternative to general anaesthetic. It is cheaper and has the potential to be more accessible. Oximetry(measurement of oxygen status) is the current gold standard in dental sedation. The main risk to the patient during sedation is a slowing of breathing due to the effects of the sedative drug. Studies from other settings where sedation is practiced suggest that an additional monitor with capnography facilitates early detection of depressed breathing. However, the results of studies from other medical settings cannot be generalised to dental sedation, because of different techniques used and the types of patients. The depth of sedation may also be vary. For dental sedation, patients remain responsive at all times and breathe for themselves. Capnography gives breath by breath information using a simple device placed close to the nose and mouth. It has been recommended by several governing medical bodies that each area of medicine, should develop its own guidelines for sedation. Therefore, there is a need to research the application of capnography for dental sedation. The proposed study will take place at a university hospital site. Patients will be randomly divided into two groups. Both groups will receive sedation in the normal way. The study group will have capnography monitoring added. The study will look for differences in breathing between the two groups. Additional information regarding other aspects of monitoring will also be obtained. The results from the proposed study may help to improve patient safety and change current practice during sedation for dentistry.

DETAILED DESCRIPTION:
Background Intravenous sedation allows procedures to be performed in dentistry, and other areas of medicine beyond the operating room. Its application in each area is tailored to the requirements of the relevant procedure, the setting and the levels of operator training and expertise. The Academy of Medical Royal Colleges emphasises that each speciality must produce its own form of guidance in the use of sedative techniques. The following definition for conscious sedation in dentistry is accepted by the General Dental Council and the Dental Sedation Teachers Group: "A technique in which the use of a drug or drugs produces a state of depression of the central nervous system enabling treatment to be carried out, but during which verbal contact with the patient is maintained throughout the period of sedation. The drugs and techniques used to provide conscious sedation for dental treatment should carry a margin of safety wide enough to render loss of consciousness unlikely". The Standing Dental Advisory Committee Guidance 2003, which remains the standard of guidance in the UK, further states: "Any technique resulting in the loss of consciousness is defined as general anaesthesia and in the UKm 'deep sedation' is considered within this category". To summarise; dental sedation lies within the range of minimal to moderate sedation on the sedation continuum i.e. conscious sedation. Deep sedation is to be avoided in this setting.

Dentists who have completed a recognised postgraduate course can practice conscious sedation independently. For intravenous sedation, dentists use a "standard" conscious sedation technique, defined as "intravenous sedation", using midazolam alone. The drug is titrated to an end-point; it is rapid in onset and possesses a short duration of action, which means that midazolam is very useful in the field of dental sedation.

The current standard of monitoring for patients is clinical monitoring, which must be supplemented by pulse oximetry and blood pressure readings. The most important side effect of midazolam is respiratory depression.

Although it is generally considered a safe practice, conscious sedation is not entirely risk-free.Ventilation (breathing) and oxygenation are related but seperate physiological processes. During the process of sedation, clinicians rely on pulse oximetry as a surrogate measure of ventilation. Capnography, a staple gold standard in general anaesthesia, is becoming an increasingly important area of interest for procedural sedation, with studies from other settings suggesting, capnography to be an effective ventilatory monitor for sedated patients.

One significant limitation of pulse oximetry is the lag time; this means that the partial pressure of oxygen may decrease significantly before the pulse oximeter signals the fall.

Reviewing the literature Previous studies on capnography for sedation are difficult to summarise. A review of the available literature has shown a relative paucity of randomised trials and no trials in the dental setting. Three trials from other settings are summarised here. Beitz et al (2012): A total of 760 patients were enrolled. Patients received 2L/min of supplemental oxygen. The intention-to-treat analysis revealed a significant reduction in the incidence of oxygen desaturation in the capnography arm in comparison with the conventional arm (38.9% vs. 53.2%). The study conclusion was that additional capnography monitoring reduces the incidence of oxygen desaturation and hypoxemia during propofol sedation for colonoscopy. Deitch et al (2010): A total of 132 patients in an emergency room setting. Hypoxia was defined as an SpO2 < 93%. The incidence of oxygen desaturation in the capnography arm in comparison with the conventional arm was 25% vs. 42%. All patients received supplemental oxygen (3L/minute). Conclusion: The addition of capnography to standard monitoring reduced the incidence of hypoxia and provided advanced warning for all hypoxic events. Qadeer et al (2009):This trial showed a significantly reduced rate of hypoxia (46% vs 69%), defined as an oximetry reading < 90% for 15 sec. There was a relatively large cohort of ASA 3 patients in the study. 147 patients received supplemental oxygen. The study conclusion was that capnography monitoring of respiratory activity improves patient safety during procedural sedation for elective endoscopy.

Waugh et al (2010) conducted a meta - analysis, the main finding being that during procedural sedation , cases of respiratory depression were 17.6 times more likely to be detected if monitored by capnography than cases not monitored by capnography ( 95% CI, 2.5-122.1).

The results from the three randomised trials and the meta-analysis cannot be generalised and extrapolated to the standard dental sedation technique because of:

1. Different patient populations The reviewed studies contain many elderly patients who are known to be more sensitive to sedative drugs and more likely to have co - morbidities. For standard dental sedation the age is less than 65 years.
2. Supplemental Oxygen In standard dental technique patients breath room air. In the reviewed studies supplemental oxygen was often administered.
3. Drugs Different drugs were used to achieve sedation in the reviewed studies e.g. Propofol and Ketamine.
4. Analgesia Local anaesthetic is employed for analgesia in dentistry. In the reviewed studies, analgesia was often achieved with the use of intravenous agents such as opioids. The synergistic effect of drugs used in combination are likely to have resulted in increased respiratory depression.
5. Desaturation (SpO2) For the standard dental sedation technique an SpO2< 95% is regarded as the threshold for early desaturation.This is a reasonable threshold in this setting where sedation is administered by a non-anaesthetist outside of the operating room. In the reviewed studies the thresholds varied. Deitch et al used a threshold < 93% and Qadeer et al. <90%.
6. Depth of sedation Varied between the studies and in some cases was beyond conscious sedation.

Aim:

The aim of this randomized, controlled study is to determine whether early intervention based upon data from capnographic monitoring reduces the incidence of arterial oxygen desaturation during midazolam sedation for dentistry.

Objectives:

1. Determine if early intervention based on capnography will influence the incidence of arterial oxygen desaturation.
2. Characterise the ETCO2, respiratory rate and SPO2 at baseline pre sedation, during sedation and post sedation.

This will be a prospective, randomised controlled trial on dental patients receiving intravenous conscious sedation with midazolam.

Goal: To determine whether use by the dental team of real - time capnography is associated with a decrease in the incidence of oxygen desaturation (hypoxia) compared with standard monitoring alone during intravenous sedation with midazolam for dentistry.

Setting and selection of participants:

Patients attending the oral surgery department and the dental theatre for sedation procedures at Cork University dentalo school and Hospital and Cork University Hospital will be prospectively invited to take part. Patients will be randomly assigned to the study group (standard monitoring and capnography) or control group (standard monitoring and blinded capnography) . The sedation team will be blinded to the randomisation choice until after enrolment. A member of staff not directly involved in the study will conduct the randomisation. There is evidence for utilising intravenous midazolam in the age group 14 to 16years (post pubertal) for dentistry. Including this age cohort ( with parental consent) will provide additional research data to add to the body of evidence. Patients will have intravenous sedation with midazolam primarily for the relief of anxiety and to help them to accept invasive procedures. The operative procedures will range from simple extractions to minor oral surgery procedures such as the removal of impacted wisdom teeth.

Pre sedation visit:

Patients will be assessed as to their suitability for sedation at a separate pre sedation visit Baseline capnography and pulse oximetry data will be collected at this visit. Patients meeting the inclusion criteria will be given written information about the study. This information will be written in lay language.

Enrolment to the study will take place at the beginning of the subsequent treatment visit for those patients who consent to take part having had time to consider the information provided about the study at the pre assessment visit. Patients will receive pre sedation instructions. Standard electronic monitoring (pulse oximetry, pulse rate and blood pressure) will be available to the clinical staff at all times. Standard dental sedation will be used according to the institutions policy and protocol. A capnostream 20 monitor ( Oridian medical, Needham, MA), using a disposable oral - nasal CO2 cannula capable of delivering oxygen, with an oral sampling port to accommodate mouth breathing will be attached to all patients. The capnostream 20 monitor displays oximetry and CO2 waveform and calculates ETCO2. The capnography monitor will be calibrated every day of the study.

Continuous recording of SpO2, Heart rate, ETCO2 and respiratory rate will be stored on a laptop computer via specialised software for post hoc analysis. In addition, clinical staff will keep paper records of the patients' age, sex, body mass index, ASA status and medical history. All patients will be assigned a code to maintain confidentiality.

Before the study, all clinicians and nursing staff will be trained in the interpretation of capnography in relation to respiratory depression including waveform interpretation. A laminated interpretation card will be attached to the monitor as a reminder. The sedation team will perform conscious sedation according to standard protocol for dental sedation. Intervention for an adverse event will be based on judgement and clinician expertise with or without capnography depending on randomisation arm. In the capnography arm,in addition to standard monitoring, changes in the shape of the capnography waveform, ETCO2 numeric changes will be considered as triggers to take measures to avoid desaturation. In the control group, capnography will be blinded by placing an opaque screen over the capnostream 20 capnographydisplay of ETCO2 values, respiratory rate and waveform. Pulse oximetry will continue to be displayed. Baseline monitoring data will be obtained for at least 2 minutes prior to the first infusion. Midazolam will be titrated at a rate of one mg per minute to an end point. Most patients are discharged 60 minutes after the last increment provided they are fit for discharge. We propose collecting study data until discharge.

All patients will receive written pre and post sedation instructions. the benzodiazepine antagonist , flumazenil will be available in the sedation suite at all times in addition to emergency drugs and equipment.

The Null hypothesis states: The study group is the same or equal to the control group in terms of hypoxemia rates i.e arterial oxygen desaturation.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anaesthesiologists (ASA) class 1 & 2 only
2. Age 14years to 65 years
3. Ability to give written informed consent

Exclusion Criteria:

1. Inability to give informed consent
2. Body Mass Index > 35 Kg/M2
3. Procedure in the upper anterior region of the mouth which prevents placement of the oral - nasal sampling device

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2013-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Arterial oxygen desaturation (SpO2 < 95%) | "participants will be followed for the duration of their sedation appointment, an expected average of one hour"
  This primary outcome measure was chosen in part because it represents a threshold point for sedation staff to stimulate patients to breathe via tactile or verbal actions.

SECONDARY OUTCOMES:
Degree of hypoxemia | "participants will be followed for the duration of their sedation appointment, an expected average of one hour
  Degree of hypoxemia; Normal (95% and above) Mild (93% to 94.99%), Moderate (90% to 92.99%) Severe hypoxemia (< 90%)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Brady, BDS MFDs, Principal Investigator — University College Cork
Locations (1):
- University College Cork, Cork, County Cork, Ireland

REFERENCES:
- [Background] implementing and ensuring safe sedation practice for healthcare procedures in adults. report of an intercollegiate working party chaired by the royal college of anaesthetists. uk academy of medical royal colleges and their faculties (2001).
- [Background] conscious sedation in the provision of dental care. report of an expert group on sedation for dentistry. standing dental advisory committee, department of health (2003)
- [Background] standards for dental professionals. U.K. general dental council (2005).
- [Background] conscious sedation in dentistry: the competent graduate: dental sedation teachers group(2000).
- [Background] standards for conscious sedation in dentistry: alternative techniques. a report from the standing committee on sedation for dentistry, faculty of dental surgery of the royal college of surgeons in england (2007)
- [Background] Beitz A, Riphaus A, Meining A, Kronshage T, Geist C, Wagenpfeil S, Weber A, Jung A, Bajbouj M, Pox C, Schneider G, Schmid RM, Wehrmann T, von Delius S. Capnographic monitoring reduces the incidence of arterial oxygen desaturation and hypoxemia during propofol sedation for colonoscopy: a randomized, controlled study (ColoCap Study). Am J Gastroenterol. 2012 Aug;107(8):1205-12. doi: 10.1038/ajg.2012.136. Epub 2012 May 29. PMID 22641306
- [Background] Deitch K, Miner J, Chudnofsky CR, Dominici P, Latta D. Does end tidal CO2 monitoring during emergency department procedural sedation and analgesia with propofol decrease the incidence of hypoxic events? A randomized, controlled trial. Ann Emerg Med. 2010 Mar;55(3):258-64. doi: 10.1016/j.annemergmed.2009.07.030. Epub 2009 Sep 24. PMID 19783324
- [Background] Qadeer MA, Vargo JJ, Dumot JA, Lopez R, Trolli PA, Stevens T, Parsi MA, Sanaka MR, Zuccaro G. Capnographic monitoring of respiratory activity improves safety of sedation for endoscopic cholangiopancreatography and ultrasonography. Gastroenterology. 2009 May;136(5):1568-76; quiz 1819-20. doi: 10.1053/j.gastro.2009.02.004. PMID 19422079
- [Background] Hart LS, Berns SD, Houck CS, Boenning DA. The value of end-tidal CO2 monitoring when comparing three methods of conscious sedation for children undergoing painful procedures in the emergency department. Pediatr Emerg Care. 1997 Jun;13(3):189-93. doi: 10.1097/00006565-199706000-00004. PMID 9220504
- [Background] Vargo JJ, Zuccaro G Jr, Dumot JA, Conwell DL, Morrow JB, Shay SS. Automated graphic assessment of respiratory activity is superior to pulse oximetry and visual assessment for the detection of early respiratory depression during therapeutic upper endoscopy. Gastrointest Endosc. 2002 Jun;55(7):826-31. doi: 10.1067/mge.2002.124208. PMID 12024135
- [Background] Tobias JD. End-tidal carbon dioxide monitoring during sedation with a combination of midazolam and ketamine for children undergoing painful, invasive procedures. Pediatr Emerg Care. 1999 Jun;15(3):173-5. doi: 10.1097/00006565-199906000-00002. PMID 10389951
- [Background] Sivilotti ML, Messenger DW, van Vlymen J, Dungey PE, Murray HE. A comparative evaluation of capnometry versus pulse oximetry during procedural sedation and analgesia on room air. CJEM. 2010 Sep;12(5):397-404. doi: 10.1017/s1481803500012549. PMID 20880431
- [Background] Miner JR, Heegaard W, Plummer D. End-tidal carbon dioxide monitoring during procedural sedation. Acad Emerg Med. 2002 Apr;9(4):275-80. doi: 10.1111/j.1553-2712.2002.tb01318.x. PMID 11927449